CLINICAL TRIAL: NCT00635453
Title: Impact of the "Ten Steps for Healthy Feeding of Children Younger Than Two Years" in Health Centers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other); Ministry of Health, Brazil (Other Government)
Responsible Party: Principal Investigator, Marcia Regina Vitolo, Professor, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: vitolo3
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Results first posted 2019-02-22 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Feeding and Eating Disorders of Childhood
Keywords: Breast Feeding; Child; Infant Nutrition Physiology; Public Health; Morbidity; Health Plan Implementation
MeSH Terms: conditions — Feeding and Eating Disorders of Childhood; Breast Feeding | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- I, Intervention (Experimental): Physicians, nurses and administrative staff of all intervention health centers participated in a training of Dietary Advice in January 2008 based on the "Ten Steps for Healthy Feeding for Brazilian Children from Birth to Two Years of Age" guideline.13 An experienced nutritionist conducted a standardized session for the health care team to outline the "Ten Steps" recommendations and strategies and to provide suggestions how best to incorporate these into the consultations. Printed materials were provided to the Health Care Centers for use by these professionals and for access to the Brazilian Ministry of Healthy Nutrition Department´s website. Health staff members received a pocket guide for use during the appointments and waiting room sessions.
  Interventions: Behavioral: Dietary Advice
- II, Control (No Intervention): Healthcare centers randomized to the non-intervention group continued their routine medical assistance without any involvement of the research team. No materials were provided to these clinics.

INTERVENTIONS:
Behavioral: Dietary Advice — The content of the dietary intervention follows the recommendations of the guidelines of the Brazilian Ministry of Health for healthy feeding of children younger then two years.
  Other Names: Infant Nutrition Programme
  Arms: I, Intervention

SUMMARY:
A cluster randomized field trial to evaluate the impact that training healthcare workers in healthy feeding practices has on the nutrition and health of children.

DETAILED DESCRIPTION:
Cluster randomized controlled trial targeting selected primary health care centers in Porto Alegre, South of Brazil, a city of 1.4 million inhabitants. The trial included health centers that provide primary care services predominantly to low-income families.Physicians, nurses and administrative staff of all intervention health centers participated in a training in January 2008 based on the "Ten Steps for Healthy Feeding for Brazilian Children from Birth to Two Years of Age" guideline.

Following staff training at the intervention sites, interviewers visited the intervention and control health centers from April to December 2008 to identify and enroll pregnant women who were in the last trimester of pregnancy. 98% of eligible pregnant women agreed to participate and answered a questionnaire about their socioeconomic status and expected due date. Addresses and telephone numbers were obtained in order to schedule subsequent home visits.

Data Collection:

Maternal interviews using structured questionnaires were conducted at baseline (during pregnancy - 2008) and at follow-up home-visits at mean child ages six months (2008/2009), 12 months (2009/2010) , three years (2011/2012) and six years (2014/2015) by field workers who were not involved in the intervention and who were unaware of the group allocations.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women in the last trimester of the gestation.

Exclusion Criteria:

* HIV-positive mothers
* congenital malformation

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 715 (Actual)
Dates: Start 2008-03-01 (Actual); Primary Completion 2010-02-28 (Actual); Study Completion 2015-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Márcia R Vitolo, Postdoctoral, Principal Investigator — Federal University of Health Sciences of Porto Alegre
Locations (1):
- The health units, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Valmorbida JL, Baratto PS, Leffa PS, Sangalli CN, Silva JA, Vitolo MR. Consumption of ultraprocessed food is associated with higher blood pressure among 6-year-old children from southern Brazil. Nutr Res. 2023 Aug;116:60-68. doi: 10.1016/j.nutres.2023.05.012. Epub 2023 May 27. PMID 37354762
- [Derived] Sangalli CN, Leffa PS, Valmorbida JL, Lumey LH, Vitolo MR. Impact of promoting healthy infant feeding practices on energy intake and anthropometric measures of children up to 6 years of age: A randomised controlled trial. J Hum Nutr Diet. 2021 Oct;34(5):771-783. doi: 10.1111/jhn.12881. Epub 2021 May 25. PMID 34034359
- [Derived] Ferreira VR, Sangalli CN, Leffa PS, Rauber F, Vitolo MR. The impact of a primary health care intervention on infant feeding practices: a cluster randomised controlled trial in Brazil. J Hum Nutr Diet. 2019 Feb;32(1):21-30. doi: 10.1111/jhn.12595. Epub 2018 Sep 4. PMID 30182376
- [Derived] Chaffee BW, Vitolo MR, Feldens CA. The Porto Alegre Early Life Nutrition and Health Study. Rev Bras Epidemiol. 2014 Dec;17(4):1015-8. doi: 10.1590/1809-4503201400040018. PMID 25388499
- [Derived] Chaffee BW, Feldens CA, Vitolo MR. Cluster-randomized trial of infant nutrition training for caries prevention. J Dent Res. 2013 Jul;92(7 Suppl):29S-36S. doi: 10.1177/0022034513484331. Epub 2013 May 20. PMID 23690364

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | I, Intervention | II, Control
Started (Pregnant woman) | 360 | 355
6 Months Assessment (Mother-Child Pairs) | 322 | 311
12 Months Assessment (Mother-Child Pairs) | 285 | 260
3 Years Assessment | 246 | 204
Completed (6 years assessment Mother-Child Pairs) | 206 | 181
Not Completed | 154 | 174

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | I, Intervention | II, Control | Total
Number analyzed (Participants) | 360 | 355 | 715
Age, Customized [Count of Participants; unit: Participants]
  < 20 years | 72 | 76 | 148
  > = 20 years | 278 | 279 | 557
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 360 | 355 | 715
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 214 | 181 | 395
  Non-White | 146 | 174 | 320
Region of Enrollment [Number; unit: participants]
  Brazil | 360 | 355 | 715

OUTCOME MEASURES:

1. Primary Outcome: Exclusive Breastfeeding at Four Months of Age
Description: Effectiveness of the nutrition advice programme will be measured comparing the number of mothers from Intervention and control groups reporting exclusively breastfeeding their infants four months after childbirth.
Time Frame: Six months after the beginning of the study
Measure: Count of Participants; unit: Participants
Arm/Group | I, Intervention | II, Control
Number analyzed (Participants) | 322 | 311
Participants | 140 | 104

2. Secondary Outcome: Number of Overweight Children at 12 Months of Age
Description: The effectiveness of the program will be evaluated by comparing number of overweight children in the intervention and control groups at 12 months of age
Time Frame: 12 months after the beginning of the study
Population: Analyzed only for participants who underwent anthropometric assessment
Measure: Count of Participants; unit: Participants
Arm/Group | I, Intervention | II, Control
Number analyzed (Participants) | 263 | 230
Participants | 124 | 112

3. Secondary Outcome: Number of Overweight Children at 3 Years of Age
Description: The effectiveness of the program will be evaluated by comparing number of overweight children in the intervention and control groups at 3 years of age
Time Frame: 3 years after the beginning of the study
Population: Analyzed only for participants who underwent anthropometric assessment and from whom post-baseline data are available.
Measure: Count of Participants; unit: Participants
Arm/Group | I, Intervention | II, Control
Number analyzed (Participants) | 238 | 216
Participants | 101 | 97

4. Secondary Outcome: Number of Overweight Children at 6 Years of Age
Description: The effectiveness of the program will be evaluated by comparing number of overweight children in the intervention and control groups at 6 years of age
Time Frame: 6 years after the beginning of the study
Population: Analyzed only for participants who underwent anthropometric assessment and from whom post-baseline data are available.
Measure: Count of Participants; unit: Participants
Arm/Group | I, Intervention | II, Control
Number analyzed (Participants) | 172 | 144
Participants | 52 | 53

5. Other Pre Specified Outcome: Food Consumption
Description: Effectiveness of a nutrition advice programme will be evaluated by comparing the food consumption differences between the intervention and control groups (nutrient and grams of non recommended food)
Time Frame: Six and twelve months, three and six years after the beginning of the study
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 years
Arm/Group | I, Intervention | II, Control
All-Cause Mortality (participants affected / at risk) | 0/360 | 0/355
Serious Adverse Events (participants affected / at risk) | 0/360 | 0/355
Other Adverse Events (participants affected / at risk) | 0/360 | 0/355

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No